CLINICAL TRIAL: NCT01116960
Title: How do Attitute About Pay for Performance Differ Among Different Anesthesia Care Provider and Over Time
Brief Title: How do Attitude About Pay for Performance Differ Among Different Anesthesia Care Provider and Over Time
Acronym: P4P
Status: Completed | Type: Observational
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Other Study IDs: 13878
Record Dates: First submitted 2010-05-03; First posted 2010-05-05 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Attitude
Keywords: P4P
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Faculty; MD: Full time Faculty members working with the Department
- CRNAs: Full time CRNAs working within the department
- Residents: Residents working within the department

SUMMARY:
The investigators hypothesize that common objections to P4P relate to potential loss of autonomy or concerns about adverse effects on patient care.

DETAILED DESCRIPTION:
We seek to establish baseline attitudes about Pay for Performance (P4P) in the OUHSC Dept of Anesthesiology and determine what differences exist between faculty, CRNAs and residents. We plan to resurvey annually to determine if attitudes change as the department implements a P4P program. We hope that by understanding the attitudes of anesthesia care providers, we can alleviate their concerns. We hope to account for their concerns as we develop and modify our P4P program. We believe that acceptance of the general idea of P4P is important if individuals are to maintain job satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* All anesthesia care providers in the department

Exclusion Criteria:

* locum faculty members and CRNAs

Ages: 24 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: anesthesia care providers
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2007-04; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Roberts, MD, Principal Investigator — University of Oklahoma
Locations (2):
- United States (2):
  - Univeristy of Oklahoma Health Sciences Center Dept. Anesthesiology, Oklahoma City, Oklahoma
  - Univeristy of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: No